CLINICAL TRIAL: NCT02826174
Title: Topical Anesthesia for Closed PKP vs Retrobulbar Anesthesia for Open-sky PKP
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Wenzhou Medical University (Other)
Responsible Party: Principal Investigator, Jinyang Li, PhD, Wenzhou Medical University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Closed PKP
Record Dates: First submitted 2016-06-21; First posted 2016-07-07 (Estimated); Last update posted 2016-07-07 (Estimated); Status verified 2016-07

CONDITIONS: Corneal Opacity; Keratitis, Herpetic; Corneal Ulcer; Corneal Dystrophies, Hereditary
MeSH Terms: conditions — Corneal Opacity; Keratitis, Herpetic; Corneal Ulcer; Corneal Dystrophies, Hereditary | interventions — Anti-Inflammatory Agents

STUDY DESIGN:
Who Masked: Participant

ARMS (4):
- closed PKP under topical anesthesia (Experimental): a closed corneal transplantation under topical anesthesia with the anterior chamber maintained
  Interventions: Procedure: closed PKP under topical anesthesia; Drug: Anti-Rejection Agents; Drug: Anti-Inflammatory Agents
- open-sky PKP under retrobulbar anesthesia (Active Comparator): an open-sky corneal transplantation under retrobulbar anesthesia
  Interventions: Procedure: open-sky PKP under retrobulbar anesthesia; Drug: Anti-Rejection Agents; Drug: Anti-Inflammatory Agents
- Anti-Rejection Agents (Other): Anti-Rejection Agents for both groups
  Interventions: Procedure: closed PKP under topical anesthesia; Procedure: open-sky PKP under retrobulbar anesthesia
- Anti-Inflammatory Agents (Other): Anti-Inflammatory Agents for both groups
  Interventions: Procedure: closed PKP under topical anesthesia; Procedure: open-sky PKP under retrobulbar anesthesia

INTERVENTIONS:
Procedure: closed PKP under topical anesthesia — a closed corneal transplantation under topical anesthesia with the anterior chamber maintained
  Arms: Anti-Inflammatory Agents; Anti-Rejection Agents; closed PKP under topical anesthesia
Procedure: open-sky PKP under retrobulbar anesthesia — an open-sky corneal transplantation under retrobulbar anesthesia
  Arms: Anti-Inflammatory Agents; Anti-Rejection Agents; open-sky PKP under retrobulbar anesthesia
Drug: Anti-Rejection Agents — Anti-Rejection Agents for both groups
  Arms: closed PKP under topical anesthesia; open-sky PKP under retrobulbar anesthesia
Drug: Anti-Inflammatory Agents — Anti-Inflammatory Agents for both groups
  Arms: closed PKP under topical anesthesia; open-sky PKP under retrobulbar anesthesia

SUMMARY:
Penetrating keratoplasty (PKP) is an open-sky surgery that fundamentally has not changed for more than 100 years. Because conventional PKP is associated with the potential for the development of devastating complications such as expulsive suprachoroidal hemorrhage and endophthalmitis, we modified the technique to one that is a closed surgery under topical anesthesia with the anterior chamber maintained to achieve favorable results. Topical anesthesia is an attractive alternative to traditional injection local anesthesia since the potentially serious complications associated with retrobulbar and peribulbar anesthesia can be avoided. The closed PKP procedure with the stable anterior chamber essentially changes the open nature of conventional PKP. The advantages, i.e., decreased surgical risks, postoperative complications, and surgical difficulties, make PKP viable in most complicated cases.

ELIGIBILITY:
Inclusion Criteria:

* active bacterial keratitis, for which ulceration progressed despite maximum antibacterial medication;
* refractory fungal keratitis that did not respond to antifungal agents;
* nonactive HSK, for which corneal opacities with or without new vessels involved the optical zone;
* ocular acid burn and thermal burn with partial limbal deficiency (50% or less) that, after more than half a year of preoperative treatment, showed reepithelialization and less than 2 quadrants limbal neovascularization.

Exclusion Criteria:

* Patients with keratolimbal allograft transplantation, total limbal stem cell deficiency secondary to ocular burns, and other ocular diseases (ie, amblyopia, age-related cataract, glaucoma, macular edema, and mac ular degeneration) were excluded.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2015-12; Primary Completion 2016-12 (Estimated); Study Completion 2016-12 (Estimated)

PRIMARY OUTCOMES:
best corrected visual acuity | preoperative
best corrected visual acuity | 1 week after PKP
best corrected visual acuity | 2 weeks after PKP
best corrected visual acuity | 1 month after PKP
best corrected visual acuity | 3 months after PKP
best corrected visual acuity | 6 months after PKP

SECONDARY OUTCOMES:
Endothelial cell density | 1 week after PKP
Endothelial cell density | 2 weeks after PKP
Endothelial cell density | 1 month after PKP
Endothelial cell density | 3 months after PKP
Endothelial cell density | 6 months after PKP

CONTACTS AND LOCATIONS:
Locations (1):
- Eye Hospital, Wenzhou Medical College, Wenzhou, Zhejiang, China

REFERENCES:
- [Background] Chen W, Ren Y, Zheng Q, Li J, Waller SG. Securing the anterior chamber in penetrating keratoplasty: an innovative surgical technique. Cornea. 2013 Sep;32(9):1291-5. doi: 10.1097/ICO.0b013e31829954c5. PMID 23860425